CLINICAL TRIAL: NCT07151612
Title: The Development of New Functions of Esculin and Digitalis Glycosides Eye Drops: A Study on the Treatment of Presbyopia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yan Gao (Other)
Responsible Party: Sponsor-Investigator, Yan Gao, Ethics Committee Contacts, Shanxi Eye Hospital
Organization: Shanxi Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SXYYLL-20240310
Record Dates: First submitted 2025-08-04; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Esculin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline solution (Placebo Comparator): The control group received an equivalent volume of sterile, preservative-free, nonirritating saline packaged in identical containers to maintain blinding.
  Interventions: Drug: Normal saline solution
- Esculin and Digitalisglycosides Eye Drops (Experimental): The treatment group received esculin and digitalis glycosides eye drops (Pharma Stulln GmbH). Patients were instructed to instill one drop in the affected eye three times daily, with strict adherence to aseptic techniques to prevent dropper-to-ocular surface contact.
  Interventions: Drug: Esculin and Digitalisglycosides Eye Drops

INTERVENTIONS:
Drug: Esculin and Digitalisglycosides Eye Drops — Interventions were performed using esculin and digitalis glycosides eye drops (Pharma Stulln GmbH). The carer instructed the patient to apply 1 drop to the affected eye three times a day and to strictly follow aseptic techniques to prevent contact of the dropper with the ocular surface. The treatment lasted for 1 month.
  Arms: Esculin and Digitalisglycosides Eye Drops
Drug: Normal saline solution — Sterile, preservative-free, and non-irritating dropper saline was used. The carer instructed the patient to apply 1 drop to the affected eye three times a day and to strictly follow aseptic techniques to prevent contact of the dropper with the ocular surface.
  Arms: Normal saline solution

SUMMARY:
Presbyopia is a condition where the eyes cannot focus a clear image on the retina when looking at nearby objects, commonly seen in people over 40 years old, which has a serious impact on people's daily work and life. However, up to now, there have been no reports in China about the approval of presbyopia treatment drugs for marketing. The theory of presbyopia regulation mechanism suggests that the accommodation of the human eye is closely related to the contraction function of the ciliary muscle. Research has found that the main components of the marketed drug, Ginkgo biloba and Digitalis glycosides eye drops, namely ginkgolide and digitalis glycosides, can act on the ciliary muscle together and effectively enhance the accommodation function of the ciliary muscle. The above results suggest that Ginkgo biloba and Digitalis glycosides eye drops may also treat presbyopia by improving the accommodation function of the ciliary muscle. However, there have been no reports on the therapeutic effect of Ginkgo biloba and Digitalis glycosides eye drops on presbyopia. Therefore, this project will, for the first time, confirm the therapeutic effect of Ginkgo biloba and Digitalis glycosides eye drops on presbyopia based on the changes in visual quality before and after treatment in the experimental group and the control group. Moreover, it will use optometry technology and optical coherence tomography (OCT) and anterior segment blood flow information to examine and analyze the accommodation function and anterior segment OCT and anterior segment blood flow information, etc., to clarify the treatment mechanism. It is hoped that the research of this project can fill the gap in the field of presbyopia drug treatment in China.

ELIGIBILITY:
Inclusion Criteria:

* Age is within the range of 40 - 55 years old.
* After mydriasis, for one eye, the refractive power is within -0.5D - 2.0D and the astigmatism is ≤ 1.0D.
* When measuring uncorrected visual acuity with a standard logarithmic visual acuity chart, the uncorrected distance visual acuity (UDVA) of both eyes is ≥ 1.25, and the uncorrected near visual acuity (UNVA) is ≤ 0.8.
* When using a slit lamp to detect cataract development according to the LOCS Ⅲ grading standard, no NO3 - NC3 or more severe lens opacity is detected; and no ocular surface diseases, visual fatigue, or any corneal diseases (such as dry eye, corneal injury, corneal opacity, keratoconus, or having undergone corneal refractive surgery, etc.) are detected.
* The subject has not used Ginkgo biloba extract dichloride eye drops within 2 weeks; has no known or suspected allergy to digitalis - like drugs; and has not used insulin, anti - anxiety drugs, antidepressants, antipsychotics, antihistamines, antispasmodics, diuretics, etc.

Exclusion Criteria:

* Age is not in the range of 40 - 55 years old.
* After mydriasis, for one eye, the refractive power is higher than 2.0D or lower than -0.5D, or the astigmatism is higher than 1.0D.
* When measuring the uncorrected distance visual acuity (UDVA) of both eyes with a standard logarithmic visual acuity chart, if the UDVA is lower than 1.25, or the uncorrected near visual acuity (UNVA) is higher than 0.8.
* When using a slit lamp to detect cataract development according to the LOCS Ⅲ grading standard, NO3 - NC3 or more severe lens opacity is detected in the lens; or ocular surface diseases, visual fatigue, or any corneal diseases (such as dry eye, corneal injury, corneal opacity, keratoconus, or having undergone corneal refractive surgery, etc.) are detected.
* The subject has used Ginkgo biloba extract dichloride eye drops within 2 weeks; has known or suspected allergy to digitalis - like drugs; or has used insulin, anti - anxiety drugs, antidepressants, antipsychotics, antihistamines, antispasmodics, diuretics, etc.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Tear film breakup time | At the beginning of the trial and two months
  The standard tear film breakup times (BUTs) was assessed by measuring the time interval between the last complete blink and the appearance of the first corneal black spot in the stained tear film, after 1% fluorescein dye was instilled into the conjunctival sac.
Dysfunctional lens index | At the beginning of the trial and two months
  Using the iTrace visual analyzer aberration analysis system for objective measurement of patients. The dysfunctional lens index (DLI) was calculated based on the data of higher-order aberrations, contrast sensitivity, and pupil diameter. The index ranged from 5.00 to 10.00.
Modulation transfer function | At the beginning of the trial and two months
  Using the iTrace visual analyzer aberration analysis system for objective measurement of patients.
Point spread function | At the beginning of the trial and two months
  Using the iTrace visual analyzer aberration analysis system for objective measurement of patients.
Corrected near visual acuity | At the beginning of the trial, one month later, and two months later
Uncorrected distance visual acuity | At the beginning of the trial, one month later, and two months later
Uncorrected intermediate visual acuity | At the beginning of the trial, one month later, and two months later
Uncorrected near visual acuity | At the beginning of the trial, one month later, and two months later
Corrected distance visual acuity | At the beginning of the trial, one month later, and two months later
Corrected intermediate visual acuity | At the beginning of the trial, one month later, and two months later
Distance-corrected intermediate visual acuity | At the beginning of the trial, one month later, and two months later
Distance-corrected near visual acuity | At the beginning of the trial, one month later, and two months later
Contrast sensitivity function | At the beginning of the trial and two months
  Contrast sensitivity (CS) measures the resolution ability of the human eye under different contrast and different spatial frequencies, which can more comprehensively evaluate the visual function of the human eye. Numerically, it is the inverse of the contrast threshold. The lower the contrast threshold of the human eye, the higher the contrast sensitivity, and the better the visual function.The patient should sit 3 meters away from this chart, wearing the best refractive correction glasses. First measure the right eye, then the left eye. The measurement sequence should be from Chart One to Chart Four, with the visual targets getting smaller from large to small. Continue until the patient cannot correctly read the two smallest visual targets on the smallest line. Try to encourage the patient to read the next smaller line of visual targets.
Total higher-order aberrations (tHOA) | At the beginning of the trial and two months
  otal higher-order aberrations (tHOA) of the whole eye within a central 3-mm optical zone was measured at baseline and after one month of treatment via an iTrace ray-tracing aberrometer (Tracey Technologies, Houston, TX, USA).The unit is root mean square (RMS)
Coma aberration | At the beginning of the trial and two months
  Coma aberration of the whole eye within a central 3-mm optical zone was measured at baseline and after one month of treatment via an iTrace ray-tracing aberrometer (Tracey Technologies, Houston, TX, USA).The unit is root mean square (RMS)
Spherical aberration | At the beginning of the trial and two months
  Spherical aberration of the whole eye within a central 3-mm optical zone was measured at baseline and after one month of treatment via an iTrace ray-tracing aberrometer (Tracey Technologies, Houston, TX, USA).The unit is root mean square (RMS)
Trefoil aberration | At the beginning of the trial and two months
  Trefoil aberration of the whole eye within a central 3-mm optical zone was measured at baseline and after one month of treatment via an iTrace ray-tracing aberrometer (Tracey Technologies, Houston, TX, USA).The unit is root mean square (RMS)

SECONDARY OUTCOMES:
Pupil diameter | At the beginning of the trial and one month later
Lens thickness | At the beginning of the trial and one month later
Anterior chamber depth | At the beginning of the trial and one month later
Lens vault height | At the beginning of the trial and one month later
Diopter | At the beginning of the trial and one month later
Diopter cylinder | At the beginning of the trial and one month later

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, Principal Investigator — Shanxi Eye Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT07151612/Prot_000.pdf
  • Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT07151612/ICF_001.pdf